CLINICAL TRIAL: NCT03746600
Title: A Telemedicine and mHealth Intervention for Reducing Alcohol Consumption Among People Living With HIV/AIDS
Brief Title: Technological Intervention for Reducing Alcohol Use Among People Living With HIV/AIDS
Acronym: TRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolyn Lauckner (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Carolyn Lauckner, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FP00008294; 1K01AA025305-01A1 (NIH)
Record Dates: First submitted 2018-09-24; First posted 2018-11-19 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV/AIDS; Alcohol Drinking
Keywords: HIV/AIDS; Alcohol Drinking; Medication Adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol Drinking; Medication Adherence | interventions — Ethanol; Economics

STUDY DESIGN:
Intervention Model Description: Randomized waitlist-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Receives the eight-week intervention, "Project TRAC: Tracking and Reducing Alcohol Consumption," immediately upon enrollment. This intervention focuses on skill building and motivational enhancement for reducing alcohol consumption.
  Interventions: Behavioral: Project TRAC: Tracking and Reducing Alcohol Consumption
- Waitlist Control Group (Other): Receives the "Project TRAC: Tracking and Reducing Alcohol Consumption" alcohol reduction intervention after an 8-week, assessment-only period. This 8-wek intervention focuses on skill building and motivational enhancement for reducing alcohol consumption.
  Interventions: Behavioral: Project TRAC: Tracking and Reducing Alcohol Consumption

INTERVENTIONS:
Behavioral: Project TRAC: Tracking and Reducing Alcohol Consumption — The TRAC intervention for people living with HIV/AIDS focuses on increasing motivation and building skills for avoiding triggers and managing situations that encourage alcohol consumption. It requires eight 30-minute sessions with a counselor using videoconferencing and mobile phones. In addition to receiving the eight sessions of intervention content, participants will complete smart phone-based self-monitoring of medication adherence and alcohol consumption, which will be discussed during intervention sessions.

SUMMARY:
While advances in medication have led to greatly improved outcomes for people living with HIV/AIDS, less than one-third of all people living with the disease are adherent enough to their medication to achieve viral suppression. Alcohol consumption has been shown to have a significant effect on HIV medication adherence, so the proposed research will aim to reduce alcohol use among people living with HIV/AIDS through a technology-driven intervention. This eight-session intervention will be delivered using a combination of videoconferencing, smart phones, and Bluetooth-enabled breathalyzers for monitoring of alcohol consumption, with an overall goal of reducing alcohol use, mitigating adherence issues, and achieving optimal prevention and treatment responses for people living with HIV/AIDS.

DETAILED DESCRIPTION:
The TRAC intervention focuses on increasing motivation and building skills for avoiding triggers and managing situations that encourage drinking. It requires eight 30-minute sessions with a counselor using videoconferencing and mobile phones. In addition to receiving the eight sessions of intervention content, participants will complete smartphone-based self-monitoring of medication adherence and alcohol consumption, which will be discussed during intervention sessions. Each day, they will be texted at two random times to complete a breathalyzer reading using a BACtrack Mobile Pro, which is sold by a company with FDA clearance and utilizes law enforcement-grade sensors for determining blood alcohol level. It connects wirelessly to phones via Bluetooth, automatically uploads readings, allows the user to view their current and past readings with a mobile app, and allows them to share their readings with counselors. At the time of the breathalyzer reading, participants will also be asked to indicate via survey how many drinks they have consumed and their medication use for the day. The surveys will be programmed using Qualtrics and accessible via a link in the reminder text message. Data analytic methods will be focused on examining effects on alcohol intake, HAART adherence, and HIV-related medical outcomes (CD4 count and viral load).If shown to be feasible, acceptable, and potentially efficacious, this intervention could have a significant impact on improving the accessibility of alcohol reduction counseling among PLWHA.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* 18 years or older
* At-risk drinker
* Currently prescribed HIV medication
* Current patient at the study recruitment site(s)

Exclusion Criteria:

* Less than 18 years old
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Lauckner, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Atlanta Veterans Health Care System, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
We will not share data due to: 1) the sensitive nature of the data (small sample size and information about HIV status of participants) and 2) the fact that these preliminary data will be used to inform a larger randomized controlled trial.

REFERENCES:
- [Derived] Lauckner C, Adatorwovor R, Taylor E, Sesenu F, Tanner T, Whitmire A, Marconi V, Kershaw T, Hansen N. The tracking and reducing alcohol consumption (TRAC) intervention for veterans living with HIV/AIDS: results from a pilot randomized waitlist-controlled trial. Addict Sci Clin Pract. 2025 Dec 3;21(1):1. doi: 10.1186/s13722-025-00631-5. PMID 41339902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for this study were recruited from the Infectious Diseases Clinic of the Atlanta Veterans Affairs Medical Center between 05/2020 and 01/2023. The first participant was enrolled in 05/2020 and the last participant was enrolled in 01/2023.
Pre-assignment Details: 50 participants were enrolled and completed the baseline assessment; 3 participants dropped out before completing any intervention sessions.
Period: Overall Study
Arm/Group | Immediate Intervention Group | Waitlist Control Group
Started | 26 | 24
Completed | 21 | 21
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — dismissed from study | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention Group | Waitlist Control Group | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.08 (11.48) | 55.79 (10.00) | 53.34 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 26 | 23 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 21 | 46
  White | 1 | 1 | 2
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Problematic Alcohol Use
Description: Alcohol Use Disorders Identification Test-C (AUDIT-C): A validated, self-report instrument assessing problematic alcohol use. For this 3-item scale, scores range from 0-12. Higher values represent greater problematic alcohol use. Change= Week 8 score - Baseline score
Time Frame: Baseline, 8-week post-test
Population: Participants who had complete data for T1 (baseline) and T2 (8-week post-test).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 21 | 20
score on a scale | -0.95 (1.50) | -1.00 (3.32)

2. Primary Outcome: Change in Daily Alcohol Consumption
Description: Single item asking how many days in the past month participants consumed alcohol. Responses range from 0-31. Change= Days reported at 8 weeks - Days reported at baseline
Time Frame: Baseline (T1), Immediate follow-up at 8 weeks (T2)
Population: Participants who had complete data for T1 (baseline) and T2 (8-week post-test)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Immediate Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 20 | 20
days | -2.95 (7.78) | -2.10 (12.48)

3. Primary Outcome: Average Percent Change in Positive Breathalyzer Readings
Description: Participants completed up to 14 breathalyzer readings/week obtained by BACTrack mobile breathalyzer. This outcome compares average % of positive breathalyzer readings (breathalyzer values > 0.00) per participant at Week 1 to Week 8. Numbers should be converted to percentages to aid in interpretation (e.g., -0.10 corresponds to a 10% decrease).
Time Frame: Week 1 and Week 8 of the active intervention period
Population: Participants who completed at least one breathalyzer reading in both Week 1 and Week 8
Measure: Mean (Standard Deviation); unit: Average percent change
Arm/Group | Immediate Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 19 | 20
Average percent change | -0.10 (0.25) | -0.07 (0.30)

4. Secondary Outcome: Percent Change in HIV/AIDS Medication Adherence
Description: Single item: Participants self-report on a scale of 0-100% how much of their HIV/AIDS medication they have taken in the previous month. Scores range from 0-100. Change = Week 8 score - Baseline score.
Time Frame: Baseline, 8-week post-test
Population: participants who completed at least one follow up questionnaire and had complete data
Measure: Mean (Standard Deviation); unit: percent change in medication adherence
Arm/Group | Immediate Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 21 | 20
percent change in medication adherence | 0 (27.71) | 1.95 (6.44)

5. Secondary Outcome: Change in CD4 Count
Description: CD4 cell count as determined by medical chart
Time Frame: Baseline, 8-week post-test, 16-week follow-up
Population: Data were not collected
Arm/Group | Immediate Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Viral Load
Description: Level of HIV virus in the month as determined by medical chart
Time Frame: Baseline, 8-week post-test, 16-week follow-up
Population: data were not collected
Arm/Group | Immediate Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change in Daily HIV/AIDS Medication Adherence
Description: % change in self-reported HIV/AIDS medication as measured via daily surveys, comparing percent of days HIV/AIDS medication was taken in Week 1 to Week 8. Numbers should be converted to percentages (i.e., a decrease of -0.01 is equivalent to a 1% decrease).
Time Frame: Week 1 and Week 8 of the active intervention period
Population: Participants who completed at least 1 daily survey during Week 1 AND during Week 8
Measure: Mean (Standard Deviation); unit: average percent change
Groups:
- Immediate Intervention Group: Received the eight-week intervention, "Project TRAC: Tracking and Reducing Alcohol Consumption," immediately upon enrollment. This intervention focuses on skill building and motivational enhancement for reducing alcohol consumption.
  Project TRAC: Tracking and Reducing Alcohol Consumption: The TRAC intervention for people living with HIV/AIDS focuses on increasing motivation and building skills for avoiding triggers and managing situations that encourage alcohol consumption. It requires eight 30-minute sessions with a counselor using videoconferencing and mobile phones. In addition to receiving the eight sessions of intervention content, participants will complete smart phone-based self-monitoring of medication adherence and alcohol consumption, which will be discussed during intervention sessions.
- Waitlist Control Group: Receives the "Project TRAC: Tracking and Reducing Alcohol Consumption" alcohol reduction intervention after an 8-week, assessment-only period. This 8-week intervention focuses on skill building and motivational enhancement for reducing alcohol consumption.
  Project TRAC: Tracking and Reducing Alcohol Consumption: The TRAC intervention for people living with HIV/AIDS focuses on increasing motivation and building skills for avoiding triggers and managing situations that encourage alcohol consumption. It requires eight 30-minute sessions with a counselor using videoconferencing and mobile phones. In addition to receiving the eight sessions of intervention content, participants will complete smart phone-based self-monitoring of medication adherence and alcohol consumption, which will be discussed during intervention sessions.
Arm/Group | Immediate Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 17 | 19
average percent change | 0.01 (0.03) | -0.02 (0.06)

8. Other Pre Specified Outcome: Change in Depressive Symptomology
Description: Patient Health Questionnaire-9 (PHQ-9). For this 9-item scale, scores range from 0-27. Higher scores indicate greater depressive symptomology.
Time Frame: Baseline, 8-week post-test, 16-week follow-up
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Anxiety Symptoms
Description: Beck Anxiety Inventory. For this 21-item scale, scores range from 0-63. Higher score indicates greater anxiety symptoms.
Time Frame: Baseline, 8-week post-test, 16-week follow-up
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Self-Reported Quality of Life
Description: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q). For this 16-item scale, raw scores range from 14-70. Scores are then converted to percentages, with higher percentages equaling greater quality of life.
Time Frame: Baseline, 8-week post-test, 16-week follow-up
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Stress
Description: Perceived Stress Scale-10. For this 10-item scale, scores range from 0-40. A higher score suggests higher perceived stress levels.
Time Frame: Baseline, 8-week post-test, 16-week follow-up
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Social Support
Description: Medical Outcomes Study Social Support Survey-12 (MOS-SSS-12). For this 12-item scale, scores range from 12-60. Higher scores suggest greater levels of social support.
Time Frame: Baseline, 8-week post-test, 16-week follow-up
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Coping Behaviors
Description: Brief COPE. This 28-item scale measures use of multiple forms of coping strategies, reflected in several subscales: Self-distraction, Active coping, Denial, Substance use, Use of emotional support, Use of instrumental support, Behavioral disengagement, Venting, Positive reframing, Planning, Humor, Acceptance, Religion, and Self-blame. Scores for each subscale range from 2-8, with higher values indicating greater use of that coping strategy.
Time Frame: Baseline, 8-week post-test, 16-week follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks (during the intervention period).
Description: The study presented minimal risk
Arm/Group | Immediate Intervention Group | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03746600/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03746600/ICF_000.pdf